CLINICAL TRIAL: NCT06631235
Title: Comparison Between Aesthetic Functional Appliances and Twin Block in Correction of Skeletal Class II: Randomized Controlled Study
Brief Title: Comparison Between Aesthetic Functional Appliances and Twin Block in Correction of Skeletal Class II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A04070240R
Record Dates: First submitted 2024-09-16; First posted 2024-10-08 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Skeletal Malocclusion
Keywords: classII; mandibular advancement; twin block

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- twin block group (Other): patient treated with twin block appliance
  Interventions: Other: orthopedic appliance
- aesthetic functional group (Experimental): patient treated with aesthetic functional appliance
  Interventions: Other: aesthetic orthopedic appliance

INTERVENTIONS:
Other: orthopedic appliance — appliances are used to correct skeletal class II due to mandibular deficiency
  Arms: twin block group
Other: aesthetic orthopedic appliance — aesthetic appliances are used to correct skeletal class II due to mandibular deficiency
  Arms: aesthetic functional group

SUMMARY:
The goal of this is to evaluate the skeletal, dental and soft tissue effects between aesthetic functional appliance and Twin block appliance in treatment of skeletal class II in ( growing male/female patients)

DETAILED DESCRIPTION:
The sample will be randomly divided into 2 equal groups according to the appliance will be used:

Group 1: Aesthetic Functional appliance Group 2: Twin block

Methods:

*Radiographs (CBCT) will be taken before starting the treatment (T1) and after obtaining Class I occlusion and normal overjet (T2) by sequential appliances.

appliances.

* Lateral cephalograms -extracted from CBCT- will be used to evaluate the effect of the two appliances.
* CBCT will be used to evaluate root resorption and bony changes in the condyle .

ELIGIBILITY:
Inclusion Criteria:

* Skeletal Class II pattern with ANB angle exceeding 6° and Wits appraisal of 2 mm or more.
* Mandibular deficiency (SNB angle less than 77°).
* Growing patients.
* No prior orthodontic intervention.
* The vertical skeletal classification shows a horizontal or neutral growth pattern.
* Overjet ≥ 8mm.

Exclusion Criteria:

* Developmental abnormalities with atypical or irregular patterns of growth and maturation.
* Any indications or manifestations, as well as any prior medical records, of Tempro-Mandibular Joint (TMJ) disorders, such as the presence of clicking, pain, limitations, or deviations.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
skeletal effects | one year
  cephalometric linear and angular measurements
dental effects | one year
  cephalometric linear and angular measurements
soft tissue effects | one year
  cephalometric linear and angular measurements

SECONDARY OUTCOMES:
root resorption | one year
  root resorption measured from CBCT

OTHER OUTCOMES:
CBCT evaluation of TMJ | one year
  adverse effects of aesthetic functional appliance on the condylar head

CONTACTS AND LOCATIONS:
Overall Officials: rana ka Abuzaid, orthodontist, Principal Investigator — Egyption orthodontic socity
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
skeletal and dental results
Supporting Information: CSR
Time Frame: 2 years
Access Criteria: mandibular advancement